CLINICAL TRIAL: NCT01705860
Title: A Long Term Follow-Up to Study 017-101-09-001: Effect of Collagenase Santyl® Ointment vs. Placebo on Healing and Scarring Characteristics of 600um Dermatome Wounds
Brief Title: Long Term Follow Up to Determine the Effects of Collagenase SANTYL Ointment on Scar Formation
Status: Completed | Type: Observational
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Other Study IDs: 017-101-09-032
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Follow up to Acute Wound Scar Study
Keywords: Collagen, collagenase, scar
MeSH Terms: conditions — Cicatrix | interventions — Collagenases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Assessment: All subjects will receive same assessments.
  Interventions: Biological: Santyl

INTERVENTIONS:
Biological: Santyl

SUMMARY:
The present study will evaluate the long term effects on scar formation for dermatome-induced skin wounds treated with Collagenase Santyl® Ointment or vehicle (white petrolatum ointment) alone. The previous study, 017-101-09-001, utilized a small, experimental, cutaneous wound to evaluate both time to complete wound closure and quality of the resulting scar when Collagenase Santyl® Ointment was used to treat the wound.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be considered qualified for enrollment if they participated in the Collagenase Santyl® Ointment Study 017 101-09-001 and provide written informed consent.
* The informed consent document must be read, signed, and dated by the suubject before conducting any study procedures or exams. In addition, the informed consent document must be signed and dated by the individual who consents the subject. A photocopy of the signed informed consent document must be provided to the subject and the original signed document placed in the subject's chart.
* Subject participated in the 017-101-09-001 study and received at least one application of a test article, whether Collagenase Santyl® Ointment or White Petrolatum.

Exclusion Criteria:

* N/A

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers who were previously treated in study 017-101-09-001 with Collagenase Santyl Ointment and Vehicle (white petrolatum ointment).
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Scar Assessment | 1 Day
  Vancouver Scar Scale assessment of dermatome wounds previously treated with Santyl Ointment or White Petrolatum

SECONDARY OUTCOMES:
Scar Quality | 1 Day
  Quality of scars over time will be assessed with the BTC-2000 instrument assessment

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint; Shai Rozen, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Dallas, Texas, United States